CLINICAL TRIAL: NCT01359397
Title: Phase II Study of Docetaxel, Oxaliplatin, Capecitabine With Bevacizumab and Trastuzumab in Case of Human Epidermal Growth Factor Receptor 2 (HER2)-Positivity in Patients With Locally Advanced or Metastatic Gastric Cancer or Adenocarcinoma of the Gastro-oesophageal Junction (B-DOCT Study)
Brief Title: Docetaxel, Oxaliplatin, Capecitabine, Bevacizumab and Trastuzumab in Patients With Locally Advanced or Metastatic Gastric Cancer
Acronym: B-DOCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: M10B-DOCT; 2010-022699-30 (EudraCT Number)
Record Dates: First submitted 2011-05-17; First posted 2011-05-24 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Gastric Cancer; Adenocarcinoma of the Gastro-oesophageal Junction
Keywords: Adenoca. stomach/gastr. Junct.
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; Capecitabine; Bevacizumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Herceptin - (Active Comparator)
  Interventions: Drug: Docetaxel, Oxaliplatin, Capecitabin, Bevacizumab
- Herceptin + (Experimental)
  Interventions: Drug: Docetaxel, Oxaliplatin, Capecitabin, Bevacizumab, Trastuzumab

INTERVENTIONS:
Drug: Docetaxel, Oxaliplatin, Capecitabin, Bevacizumab — Her2 - patients only
  Arms: Herceptin -
Drug: Docetaxel, Oxaliplatin, Capecitabin, Bevacizumab, Trastuzumab — for Her2 + patients only
  Arms: Herceptin +

SUMMARY:
Background: It is estimated that in the Netherlands each year approximately 900 patients with gastric cancer or adenocarcinoma of the gastro-oesophageal junction are candidates for chemotherapy. Randomized studies comparing chemotherapy versus best supportive care have shown that survival and quality of life are prolonged with chemotherapy. However, no chemotherapy regimen is clearly superior with regard to prolongation of survival. Therefore, tolerability of treatment and ease of administration (outpatient compared to inpatient) are important considerations for the development of novel treatment schedules. Study design: This is an open-label, multicentre, phase II trial designed to evaluate the efficacy and safety of bevacizumab in combination with docetaxel, oxaliplatin and capecitabine chemotherapy (B-DOC) as first-line therapy in patients with inoperable locally advanced or recurrent and/or metastatic adenocarcinoma of the stomach or gastro-oesophageal junction. In case of HER2 positive inoperable locally advanced or recurrent and/or metastatic adenocarcinoma of the stomach or gastro-oesophageal junction trastuzumab is added to this regimen (B-DOCT).

Study Endpoints:

Primary endpoint Progression free survival defined as the time measured from B-DOCT study, Protocol version 3.0 dated January 18, 2011 Page 5 / 60 the day of registration to first progression or death. Secondary endpoints Toxicity Overall survival, defined as the time from registration to death Response rate defined as the percentage of partial and complete responses Duration of response defined as time from response to first progression Translational research on pharmacogenomic and biological factors that may predict treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the stomach or gastro-oesophageal junction with inoperable locally advanced or recurrent and/or metastatic disease not amenable to curative therapy.
2. Measurable disease, according to the Response Evaluation Criteria in Solid Tumours (RECIST), assessed using imaging techniques (CT or MRI)
3. ECOG Performance status 0, 1 or 2 (see Appendix 2)
4. Life expectancy of at least 3 months
5. Male or female age ≥ 18 years.
6. Signed informed consent.
7. Assessment of HER2 status (primary tumour or metastasis) by the central laboratory prior to initiation of study treatment (see section 9.1)
8. Able to swallow and retain oral medication.
9. LVEF ≥ 50% assessed by multigated radionucleotide angiography (MUGA) or cardiac ultrasound.

Exclusion Criteria:

Any of the following will exclude the patient from the study:

1. Previous chemotherapy for advanced/metastatic disease (prior peri-operative chemotherapy is allowed if at least 6 months has elapsed between completion of this therapy and enrolment into the study).
2. Previous radiotherapy on the abdomen.
3. Other malignancy within the last 5 years, except for carcinoma in situ of the cervix, or basal cell carcinoma.
4. Patients with active (significant or uncontrolled) gastrointestinal bleeding.
5. Residual relevant toxicity resulting from previous therapy (with the exception of alopecia), e.g. neurological toxicity ≥ grade 2 NCI-CTCAE.
6. Creatinin clearance <50 mL/min.
7. Neutrophil count <1.5 × 109/L, or platelet count <100 × 109/L.
8. Serum bilirubin >1.5 × upper limit of normal (ULN); or, AST or ALT >2.5 × ULN (or >5 × ULN in patients with liver metastases); or, alkaline phosphatase >2.5 × ULN (or >5 × ULN in patients with liver metastases, or >10 × ULN in patients with bone but no liver metastases); or, albumin <25 g/L.
9. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
10. History of documented congestive heart failure; angina pectoris requiring medication; evidence of transmural myocardial infarction on ECG; poorly controlled hypertension (systolic BP >180 mmHg or diastolic BP >100 mmHg); clinically significant valvular heart disease; or high risk uncontrollable arrhythmias.
11. Patients with dyspnoea at rest due to complications of advanced malignancy or other disease, or who require supportive oxygen therapy.
12. Patients receiving chronic or high dose corticosteroid therapy. (Inhaled steroids and short courses of oral steroids for anti-emesis or as an appetite stimulant are allowed).
13. Major surgery within 4 weeks of start of study treatment; serious or not healing wound.
14. Known hypersensitivity to any of the study drugs, Chinese hamster ovary cell products or other murine or human recombinant antibodies.
15. History or clinical evidence of brain metastases.
16. Serious uncontrolled systemic intercurrent illness, e.g. infections or poorly controlled diabetes.
17. Positive serum pregnancy test in women of childbearing potential.
18. Subjects with reproductive potential not willing to use an effective method of contraception.
19. Any investigational drug treatment within 4 weeks of start of study treatment.
20. Radiotherapy within 4 weeks of start of study treatment (2 week interval allowed if palliative radiotherapy given to bone metastastic site peripherally and patient recovered from any acute toxicity)
21. Arterial thrombosis; cerebrovascular accident within 6 months prior to study enrolment.
22. Therapeutic use of oral coumarin-derived or LMWH anticoagulants or NSAIDs.
23. Continuous use of immunosuppressive agents (for the use of corticosteroids see also #12).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2011-03; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Patients will be followed for an average period of 1 year
  the time measured from the day of registration to first progression or death

SECONDARY OUTCOMES:
Number of Participants with Serious Adverse Events as a Measure of Safety and Tolerability | Patients will be followed for an average period of 1 year
  Toxicity will be evaluated during/after every course. Patients having received ≥1 treatment doses are evaluable for toxicity. Evaluation will be performed on the safety population (having received treatment). Clinical and laboratory toxicity will be graded according to NCI common toxicity criteria, version 4.0.
Overall survival | 12 months
  defined as the time from registration to death Response rate defined as the percentage of partial and complete responses Duration of response defined as time from response to first progression

CONTACTS AND LOCATIONS:
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

REFERENCES:
- See also: Related Info — http://www.dccg.nl/dccg-trials/b-doct/